CLINICAL TRIAL: NCT00140881
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Determine the Effect of Montelukast Sodium as an Episode Modifier in the Treatment of Infrequent Episodic Asthma in Children
Brief Title: A Study to Determine the Effect of Montelukast Sodium as an Episode Modifier in the Treatment of Infrequent Episodic Asthma in Children (0476-165)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-165; 2005_055
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2024-08-14 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

INTERVENTIONS:
Drug: MK0476; montelukast sodium
Drug: Comparator: placebo

SUMMARY:
A 53-week study to determine the effect of montelukast sodium when given to children (with infrequent episodic asthma) at the earliest symptoms of an acute episode of asthma.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 2 and 14 who have infrequent episodic asthma.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2000-06-01 (Actual); Primary Completion 2003-02-14 (Actual); Study Completion 2003-02-14 (Actual)

PRIMARY OUTCOMES:
Composite unscheduled acute health care resource utilisation (specific for asthma; unscheduled visits, GP attendance, ED attendance and hospital admission).

SECONDARY OUTCOMES:
Parent/caregiver QOL endpoints.
The safety and tolerability of montelukast when use as an episode modifier.
The duration and severity of the episode assessed by the parent/caregiver symptom score and the use of b-agonist and oral corticosteroid.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Robertson CF, Price D, Henry R, Mellis C, Glasgow N, Fitzgerald D, Lee AJ, Turner J, Sant M. Short-course montelukast for intermittent asthma in children: a randomized controlled trial. Am J Respir Crit Care Med. 2007 Feb 15;175(4):323-9. doi: 10.1164/rccm.200510-1546OC. Epub 2006 Nov 16. PMID 17110643